CLINICAL TRIAL: NCT00236977
Title: Comparison of the Safety and Efficacy of Intravenous Iron Versus Oral Iron in Chronic Renal Failure Subjects With Anemia
Brief Title: Comparison of Safety and Efficacy of Intravenous Iron Versus Oral Iron in Chronic Renal Failure Subjects With Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Marc L. Tokars, Luitpold Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VEN03027
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Anemia
Keywords: CKD; iron; anemia
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated; ferrous sulfate; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venofer (Experimental): iron sucrose injection
  Interventions: Drug: Venofer
- Ferrous Sulfate (Active Comparator): oral iron
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Venofer — iron sucrose injection; 500 mg intravenous (IV) infusion administered over 3.5-4 hours on Days 0 and 14, or 200 mg injections administered over 2-5 minutes on 5 different occasions from Day 0 to Day 14.
  Other Names: iron sucrose tablets
  Arms: Venofer
Drug: Ferrous Sulfate — oral iron tablets; 325 mg three times a day orally for 56 days
  Other Names: Oral Iron Tablets
  Arms: Ferrous Sulfate

SUMMARY:
To assess the safety and efficacy of two forms of iron therapy for the treatment of anemia in non-dialysis dependent, chronic renal failure in patients receiving or not receiving erythropoietin.

DETAILED DESCRIPTION:
The intent of this study was to assess the safety and efficacy of two forms of iron therapy for the treatment of anemia in non-dialysis dependent, chronic renal failure patients receiving or not receiving erythropoietin. After an extensive enrollment period, patients were randomized to receive oral iron (ferrous sulfate, 325mg three times daily (TID) for 56 days) or IV iron sucrose (total 1000mg, 500mg X 2 OR 200mg X 5 within two weeks). Erythropoietin schedule was to remain unchanged during the 56 day study.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin < or = 11.5 gm/dL
* Stable dose or not receiving EPO
* Renal Anemia

Exclusion Criteria:

* IV iron with last 6 months
* Chronic infection, malignancy,major surgery within last month
* Blood Transfusion with last two months
* Significant blood loss within last 3 months
* Concomitant sever diseases of the liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2003-08; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Falone, MD, Study Director — American Regent, Inc.
Locations (1):
- Luitpold Pharmaceuticals, Valley Forge, Pennsylvania, United States

REFERENCES:
- [Result] Van Wyck DB, Roppolo M, Martinez CO, Mazey RM, McMurray S; United States Iron Sucrose (Venofer) Clinical Trials Group. A randomized, controlled trial comparing IV iron sucrose to oral iron in anemic patients with nondialysis-dependent CKD. Kidney Int. 2005 Dec;68(6):2846-56. doi: 10.1111/j.1523-1755.2005.00758.x. PMID 16316362

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: August 2003 to October 2004. Locations: Hospitals, Medical Clinics
Pre-assignment Details: Eligibility requirements: Serum Transferrin Saturation (TSAT) <= to 25%, Ferritin <= to 300 ng/mL, and no iron following enrollment. At randomization subjects were stratified by gender, hemoglobin (Hgb) levels (< or = to 9.0 g/dL, 9.1 - 10.0 g/dL, 10.1 - 11.0 g/dL), and erythropoietin use.
Period: Overall Study
Arm/Group | Venofer | Ferrous Sulfate
Started | 91 | 91
Completed | 70 | 72
Not Completed | 21 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venofer | Ferrous Sulfate | Total
Number analyzed (Participants) | 91 | 91 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 43 | 92
  >=65 years | 42 | 48 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 64 | 126
  Male | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Patients With an Increase in Hemoglobin >= 1gm/dL.
Time Frame: Change from Baseline up to Day 56
Population: Intent to Treat (ITT) population exclusions: Venofer - 12 subjects excluded; Ferrous Sulfate - 9 subjects excluded; due to either no post-baseline efficacy data, or unstable use of erythropoietin during the eight weeks prior to randomization.
Measure: Number; unit: participants
Arm/Group | Venofer | Ferrous Sulfate
Number analyzed (Participants) | 79 | 82
participants | 35 | 23

2. Secondary Outcome: Number of Subjects With a Clinical Response
Description: Clinical Response (change in Hemoblobin (Hgb) >= 1gm/dL and change in ferritin >= 160ng/ml)
Time Frame: Change from Baseline up to Day 56
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Venofer | Ferrous Sulfate
Number analyzed (Participants) | 79 | 82
participants | 31 | 1

3. Secondary Outcome: Highest Change From Baseline in Hemoglobin (g/dL) up to Day 56
Time Frame: Change from Baseline up to Day 56
Population: Only subjects who completed the study from the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Venofer | Ferrous Sulfate
Number analyzed (Participants) | 67 | 65
g/dL | 1.1 (.94) | .8 (.78)

4. Secondary Outcome: Highest Change From Baseline in Ferritin (ng/mL) up to Day 56
Time Frame: Change from Baseline up to Day 56
Population: Only subjects who completed the study from the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Venofer | Ferrous Sulfate
Number analyzed (Participants) | 67 | 65
ng/mL | 391.7 (213.19) | 45 (52.19)

5. Secondary Outcome: Mean Change in Ferritin (ng/mL) From Baseline to Day 56
Time Frame: Change from Baseline at Day 56
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Venofer | Ferrous Sulfate
Number analyzed (Participants) | 79 | 82
ng/mL | 230 (138.2) | 30 (54.63)

6. Secondary Outcome: Mean Change From Baseline in Serum Transferrin Saturation (TSAT) (%) at Day 56
Time Frame: Change from Baseline at Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Venofer | Ferrous Sulfate
Number analyzed (Participants) | 79 | 82
percentage of change | 8.5 (8.31) | 5.5 (9.14)

7. Secondary Outcome: Mean Change From Baseline in Hemoglobin (g/dL) at Day 56
Time Frame: Change from Baseline at Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Venofer | Ferrous Sulfate
Number analyzed (Participants) | 79 | 82
g/dL | .7 (.94) | .3 (.90)

ADVERSE EVENTS:
Time Frame: 1 year and 2 months
Arm/Group | Venofer | Ferrous Sulfate
Serious Adverse Events (participants affected / at risk) | 10/91 | 6/91
Other Adverse Events (participants affected / at risk) | 37/91 | 42/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venofer (N=91) | Ferrous Sulfate (N=91)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fracture reduction (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension NOS (Vascular disorders) | 2 (2) | 0 (0)
Intraoperative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lobar pneumonia NOS (Infections and infestations) | 1 (1) | 0 (0)
Mental status changes (General disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia NOS (Infections and infestations) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis NOS (Infections and infestations) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venofer (N=91) | Ferrous Sulfate (N=91)
Constipation (Gastrointestinal disorders) | 5 (5) | 11 (11)
Diarrhea NOS (Gastrointestinal disorders) | 5 (5) | 9 (9)
Dizziness (Nervous system disorders) | 5 (6) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 7 (12) | 0 (0)
Fatigue (General disorders) | 3 (4) | 6 (6)
Fecal Occult Blood Positive (Investigations) | 2 (2) | 5 (7)
Hypertension NOS (Vascular disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 9 (10)
Oedema NOS (General disorders) | 4 (4) | 8 (8)
Oedema peripheral (General disorders) | 7 (8) | 2 (2)
Urinary Tract Infection NOS (Infections and infestations) | 1 (1) | 6 (6)
Vomiting NOS (Gastrointestinal disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less